CLINICAL TRIAL: NCT05201430
Title: Neoadjuvant FOLFOXIRI Chemotherapy Versus CapeOX Chemotherapy for Local Advanced Rectal Cancer: An Open Label Randomized Controlled Phase III Trial
Brief Title: Neoadjuvant FOLFOXIRI Versus CapeOX Chemotherapy for Local Advanced Rectal Cancer
Acronym: RCNAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, Professor, Chief of Department of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2108240-5
Record Dates: First submitted 2021-12-04; First posted 2022-01-21 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant chemotherapy; Locally advanced rectal cancer; FOLFOXIRI; CapeOX
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Fluorouracil; Oxaliplatin; Irinotecan; Surgical Procedures, Operative; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: FOLFOXIRI (Experimental): Neoadjuvant chemotherapy with 3-4 cycles of FOLFOXIRI regimen, followed by surgery
  Interventions: Drug: FOLFOXIRI
- B: CapeOX (Experimental): Neoadjuvant chemotherapy with 2-3 cycles of CapeOX regimen, followed by surgery
  Interventions: Drug: CapeOX

INTERVENTIONS:
Drug: FOLFOXIRI — irinotecan* 165 mg/m² iv continue for 1.5 hours, D1 oxaliplatin 85 mg/m² iv continue for 2 hours, D1 leucovorin 400 mg/m² iv continue for 2 hours, D1 5-FU 2400~3200 mg/m² cont. inf. 48h, D1 repeat every 2 weeks (Q2W)
  Other Names: 5-Fu; Oxaliplatin; Irinotecan; Surgery
  Arms: A: FOLFOXIRI
Drug: CapeOX — oxaliplatin 130 mg/m2 iv continue for 2 hours, D1 capecitabine 1000mg/m2/d PO Bid, once every morning and evening D1-14 repeat every 3 weeks (Q3W)
  Other Names: Capecitabine; Oxaliplatin; Surgery
  Arms: B: CapeOX

SUMMARY:
This is a phase III randomized controlled trial comparing the efficacy and safety of FOLFOXIRI versus CapeOX as neoadjuvant regimen in treating patients with middle and upper locally advanced (MRI T3-4 or N+) rectal cancer. This study aims to optimize the neoadjuvant therapy for patients with anus-preserving resectable locally advanced rectal cancer, so as to improve the prognosis of them. It remains unclear about whether FOLFOXIRI or CapeOX neoadjuvant chemotherapy is more effective for locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* MRI evaluated of T3-4 or N+ rectal cancer;
* Pathologically diagnosed of rectal adenocarcinoma;
* 18 to 75 years old;
* Distance from lower margin of tumor to anus <15 cm and suitable for anus-preserving resection;
* Tumor amenable to radical resection;
* Treatment-na?ve patients with no previous systemic chemotherapy, radiotherapy or local excision for treating rectal cancer;
* Laboratory requirements conducted within 7 days of starting study treatment: Neutrophil count ≥ 1.5×10^9/L, Platelet count ≥ 100×10^9 /L, Hemoglobin ≥ 80 g/L, Serum bilirubin ≤ 24umol/L, Alanine aminotransferase and aspartate aminotransferase ≤ 60 U/L, Serum creatinine ≤ 110 umol/L;
* Be capable to receive a surgery;
* No second tumor at present or in the past 5 years, except skin basal cell carcinoma, skin squamous cell carcinoma, or any in situ cancer;
* No previous systemic chemotherapy for treating colorectal cancer;
* Life expectancy of more than 3 months;
* No current pregnancy or breast-feeding, and subjects at childbearing age shall take method of contraception;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1;
* Be willing and able to understand the study and to provide written informed consent.

Exclusion Criteria:

* End-stage cachexia patients;
* Cardiopulmonary dysfunction or liver and kidney dysfunction, and unable to tolerate chemotherapy or surgery;
* Metastatic carcinoma;
* Incomplete or complete intestinal obstruction;
* Known to be allergic to capecitabine, 5-Fu, oxaliplatin or irinotecan;
* Pregnant or lactating women; or women who have fertility but have not taken at taken adequate contraceptive measures;
* Have vital organ failure or other severe diseases, including but not limited to coronary heart disease, cardiovascular diseases, or myocardial infarction within 12 months before being included; severe neurological or psychiatric historysevere infection; active disseminated intravascular coagulation; active hepatitis, severe coagulation disorder patients;
* History of other malignancy within the past 5 years except effectively treated skin basal cell carcinoma, skin squamous cell carcinoma, or any in situ cancer;
* Serious organic disease including but not limited to heart, kidney, brain, and lung.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years
  Defined as the length of time from the date of randomization until the first documented date of progression or death from any cause, whichever comes first. Compare 3-year disease free survival in patients with locally advanced rectal cancer treated with either FOLFOXIRI or CapeOX neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
pathologic complete response rate | 1 year
  Defined as the ratio of patients with pathologic TRG 0
major pathologic response rate | 1 year
  Defined as the ratio of patients with pathologic TRG 0 or 1
objective response rate | 1 year
  Defined as the ratio of patients with MRI-TRG 1, 2 or 3
local recurrence rate | 3 years
  Defined as the ratio of patients with local recurrence within 3 years.
overall survival | 5 years
  Defined as the length of time from randomization date until the date of death from any cause.
quality of life as assessed by EORTC QOL-C30 | 3 years
  Quality of life after neoadjuvant chemotherapy is assessed by questionaires EORTC QOL-C30 version 3
quality of life as assessed by EORTC QOL-CR29 | 3 years
  Quality of life after neoadjuvant chemotherapy is assessed by questionaires EORTC QOL-CR29.
adverse event | 1 year
  Number of patients with adverse events and severity according to NCI CTC 5.0 after neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Xu, Principal Investigator — Fudan University
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Caner Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Proper legal IPD will be shared when publishing articles.